CLINICAL TRIAL: NCT00047476
Title: Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of d-MPH in the Treatment of Fatigue and Neurobehavioral Impairment Related to Chemotherapy in Adult Cancer Patients
Brief Title: D-MPH in the Treatment of Fatigue and Neurobehavioral Function Related to Chemotherapy in Adult Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Organization: Celgene (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: d-MPH-COG-002; NCT00052533 (obsolete NCT alias)
Record Dates: First submitted 2002-10-08; First posted 2002-10-09 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-05

CONDITIONS: Fatigue; Neoplasms
Keywords: neurobehavioral function; chemobrain; chemo brain; fatigue; memory loss; exhausted; trouble concentrating
MeSH Terms: conditions — Fatigue; Neoplasms; Chemotherapy-Related Cognitive Impairment; Memory Disorders

INTERVENTIONS:
Drug: dexmethylphenidate(d-mph)

SUMMARY:
To evaluate the efficacy of dexmethylphenidate (d-MPH) in the treatment of chemotherapy-related fatigue in adult cancer subjects.

ELIGIBILITY:
* Diagnosis of cancer, excluding primary or metastatic brain tumors.
* Treated with a minimum of four cycles of a cytotoxic chemotherapy, the last chemotherapy treatment must have been completed at least 2 months prior to study entry.
* Physical/neurological examination consistent with the absence of a focal neurological deficit
* Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).
* Subjects must be able to adhere to the protocol requirements.
* Subjects must understand and voluntarily sign an informed consent document.
* Subjects must be a native English speaker or fluent in English, and have at least an eighth grade education.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2002-06; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Cooper Green Hospital, Jefferson Clinic, Birmingham, Alabama
  - University of Alabama Palliative Care Institute, Birmingham, Alabama
  - Peak Performance Wellness, Flagstaff, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - California Cancer Care Inc, Greenbrae, California
  - Clinical Trials and Research Associates, Montebello, California
  - Comprehensive Cancer Centers of the Desert, Palm Springs, California
  - Comprehensive Cancer Center, Boca Raton, Florida
  - Osler Clinical Research/Osler Medical Inc, Melbourne, Florida
  - University of Miami, Sylvester Cancer Research Center, Miami, Florida
  - Cancer Research Network Inc, Plantation, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Markey Cancer Center, Lexington, Kentucky
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Beth Israel Cancer Center, New York, New York
  - Gynecologic Oncology Associates and Development LLC, Greenville, South Carolina
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Northwest Medical Specialists, PLLC, Tacoma, Washington
  - UW Comprehensive Cancer Center, Madison, Wisconsin